CLINICAL TRIAL: NCT02691871
Title: A Phase I, Open-label, Dose-escalation Study of Apatinib in Combination With Docetaxel as 2nd Line Treatment in Patients With Advanced Lung Adenocarcinoma Harboring Wild-type Epidermal Growth Factor Receptor (EGFR)
Brief Title: Apatinib Plus Docetaxel as 2nd Line Treatment in Patients With Advanced Lung Adenocarcinoma Harboring Wild-type EGFR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jie Wang, Chairman, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-L301
Record Dates: First submitted 2016-02-03; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — apatinib; Docetaxel

ARMS (1):
- Apatinib + Docetaxel (Experimental): Low, medium or high dose of Apatinib (days 3-19, q3w) and Docetaxel (60 mg/m2, day 1, q3w)
  Interventions: Drug: Apatinib (250 mg/d) + Docetaxel (60 mg/m2); Drug: Apatinib (500 mg/d) + Docetaxel (60 mg/m2); Drug: Apatinib (750 mg/d) + Docetaxel (60 mg/m2)

INTERVENTIONS:
Drug: Apatinib (250 mg/d) + Docetaxel (60 mg/m2)
Drug: Apatinib (500 mg/d) + Docetaxel (60 mg/m2)
Drug: Apatinib (750 mg/d) + Docetaxel (60 mg/m2)

SUMMARY:
The purpose of this study is to confirm the safety of Apatinib at a dose level up to 750 mg/d with standard therapy of docetaxel (60 mg/m²) in advanced lung adenocarcinoma patients harboring wild-type EGFR after failure of first line chemotherapy and to determine the recommended dose for the Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 65 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1;
3. Life expectancy of more than 12 weeks;
4. At least one measurable lesion according to RECIST 1.1 which has not received radiotherapy =< 3 months;
5. Histologically/cytologically confirmed advanced/metastatic lung adenocarcinoma of stage IV with documented wild-type EGFR;
6. Patients with one prior platinum-containing chemotherapy. In case of recurrent disease, one additional prior regimen is allowed for adjuvant and/or neoadjuvant therapy.
7. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 100×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1×ULN, Cr clearance ≥ 50 mL/min, INR < 1.5 or PT < ULN+4s or APTT < 1.5×ULN, proteinuria < (++) or urinary protein ≤ 1.0 g/24 hrs;
8. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
9. Signed informed consent.

Exclusion Criteria:

1. Accumulation of coelomic fluid (e.g. pleural effusion, ascites fluid, cardiac effusion) requiring treatment;
2. Other malignancy within the past five years other than basal cell skin cancer, or carcinoma in situ of the cervix;
3. Factors affecting the oral medication (e.g. inability to swallow, chronic diarrhea and intestinal obstruction);
4. Major injuries and/or surgery =< 4 weeks prior to registration with incomplete wound healing. Patients who have received radiotherapy (except local palliative radiotherapy), chemotherapy, molecular targeted therapy =< 3 weeks, or nitrosoureas/mitomycin chemotherapy =< 6 weeks prior to registration;
5. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
6. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to NYHA criteria or echocardiography check: LVEF<50%;
7. History of clinically significant haemoptysis =< 2 months (more than half of one tea spoon of fresh blood per day) prior to registration. Coagulation disfunction, hemorrhagic tendency or receiving anticoagulant therapy;
8. History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, bleeding ulcer, occult blood ≥ (++), and vasculitis) =< 3 months prior to randomization;
9. Patients who have active brain metastases or leptomeningeal disease. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation ending at least 3 weeks prior to randomization, or after surgical resection performed at least 3 weeks prior to randomization. No evidence of Grade greater than or equal to 1 CNS hemorrhage based on pretreatment CT or MRI scan;
10. Centrally located tumors of local invasion of major blood vessels, or distinct interstitial lung disease by the chest radiographic findings (CT or MRI);
11. Treatment with other investigational drugs or other anti-cancer therapy;
12. Previous therapy with other VEGFR inhibitors (other than bevacizumab);
13. Previous therapy with docetaxel =< 6 months prior to registration;
14. Treatment in another investigational trial =< 4 weeks prior to registration;
15. Any contraindications for therapy with docetaxel. History of severe hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80 (Tween 80). History of hypersensitivity to apatinib and/or the excipients of the trial drugs;
16. Active or chronic hepatitis C and/or B infection, or other active uncontrolled infection;
17. History of immunodeficiency disease (including HIV positive), concurrent acquired or congenital immunodeficiency syndrome, or history of organ transplantation;
18. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to registration;
19. History of arterial or venous thromboembolic events (e.g. CVA, DVT and pulmonary embolism) =< 12 months prior to randomization;
20. Administration of strong/potent cytochrome P450 (CYP)3A4 inhibitors within 7 days, or inducers within 12 days;
21. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study;
22. History of mental diseases;
23. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Apatinib in combination with Docetaxel (60 mg/m2) | During the first treatment course, up to 3 weeks
Number of Participants Experienced Dose Limited Toxicity (DLT) in Combination Therapy of Apatinib and Docetaxel | During the first treatment course, up to 3 weeks

SECONDARY OUTCOMES:
Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 for All Courses | Between the first administration of Docetaxel and 28 days after last administration of Apatinib, up to 1 year
Objective Response Rate (ORR) | Every 6 weeks from the first treatment course, up to 1 year
Progression-free Survival (PFS) | Every 6 weeks from the first treatment course, up to 2 year